CLINICAL TRIAL: NCT04728594
Title: Evaluation of an Email Intervention Promoting COVID-19 Vaccination Among Healthcare Workers
Brief Title: Emails Promoting COVID-19 Vaccination Among Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Michelle N. Meyer, Faculty Co-Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0128
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Vaccination Refusal; Communication
Keywords: Immunization; Persuasive Communication; Electronic Mail; Economics, Behavioral; Psychology
MeSH Terms: conditions — Vaccination Refusal; Communication; Behavior | interventions — Cognitive Restructuring

STUDY DESIGN:
Intervention Model Description: 1 x 3 design
Who Masked: Participant, Care Provider
Masking Description: Participants will not know what group they are in. The relevant care provider (either their primary care provider or provider administering the vaccine) will not know about this study or assignment into groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delayed Contact (No Intervention): This group will not receive an email for at least two days.
- Social Proof (Experimental): This group will receive an email that points out that vaccine availability for employees will soon be limited. It also emphasizes how many fellow health care workers have been vaccinated. Seeing the behaviors of other people might encourage recipients to copy that behavior.
  Interventions: Behavioral: Social Proof; Behavioral: Scarcity Message
- Reframing Side Effects and Adverse Reactions (Experimental): This group will receive an email that points out that vaccine availability for employees will soon be limited. It also addresses concerns about the side effects and adverse reactions of the vaccine. Due to potentially overblown concerns about the vaccine caused by the salience of side effects in the (social) media, the email attempts to reframe the risks by explicitly noting the small possibility of being affected by serious side effects and by contrasting that to the more severe effects of COVID-19. As a result of this reframing, recipients might recalibrate their perception of risks and benefits and opt for vaccination.
  Interventions: Behavioral: Reframing; Behavioral: Scarcity Message

INTERVENTIONS:
Behavioral: Social Proof — Email
  Arms: Social Proof
Behavioral: Reframing — Email
  Arms: Reframing Side Effects and Adverse Reactions
Behavioral: Scarcity Message — Email
  Arms: Reframing Side Effects and Adverse Reactions; Social Proof

SUMMARY:
In this evaluation, two versions of emails will be sent to Geisinger employees who have not been vaccinated against COVID-19. A delayed-contact control group will be emailed after a delay of at least two days. The researchers hypothesize that either of the emails - which use content informed by behavioral nudge theory - will lead to more COVID-19 vaccinations than the delayed-contact control group.

DETAILED DESCRIPTION:
The researchers aim to evaluate the effectiveness of email reminders in promoting COVID-19 vaccinations among Geisinger employees. The project will compare two emails, which will vary in the subject line and email content. Both emails will test different approaches that draw from principles in behavioral science: social proof, reframing, and scarcity. Employees receiving these emails will be compared with employees in a delayed-contact group, who will not receive emails. Employees in the control group will later receive one of the emails.The responses to the emails will help determine the communications later sent to the control group.

All emails will ask recipients if they want to receive a COVID-19 vaccination. If they click on a hyperlink indicating yes, they will be forwarded to an online registration and scheduling homepage. If they click on a hyperlink indicating no, they will be forwarded to an online questionnaire surveying people about their main reason for declining the vaccine at this time. The questionnaire will automatically present information intended to assuage the specific concern that people endorse, followed by a hyperlink to the scheduling site.

The data will be analyzed with logistic regression models with the control group as the reference group, to compare the two email conditions versus the control group. This set of analyses will only be conducted for scheduling a vaccination appointment as opposed to email engagement outcomes (e.g., number of emails opened), which will not be applicable for the control group. A second set of logistic regression models predicting scheduling a vaccination appointment and email engagement will also be run, comparing the two email conditions against each other. The data will be examined two days later (to help decide which email to send to the delayed-control group) and four days later (when the policy for employee vaccination will change, making the content of the email irrelevant).

Update: The researchers looked at 3 days of data - as the emails to the delayed contact group were only sent at that time - and 4 days of data when the policy for employee vaccinations changed.

ELIGIBILITY:
Inclusion Criteria:

* Employees at Geisinger Health System who have not gotten a COVID-19 vaccination

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9566 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Meyer, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

REFERENCES:
- [Derived] Santos HC, Goren A, Chabris CF, Meyer MN. Effect of Targeted Behavioral Science Messages on COVID-19 Vaccination Registration Among Employees of a Large Health System: A Randomized Trial. JAMA Netw Open. 2021 Jul 1;4(7):e2118702. doi: 10.1001/jamanetworkopen.2021.18702. PMID 34319359

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delayed Contact | Social Proof | Reframing Side Effects and Adverse Reactions
Started (Participants who were sent an email.) | 3178 (The number of participants who were sent a follow up email (delayed, three days after the other two arms) was used to see how many started.) | 3198 | 3190
Completed (Participants who were sent an email were also considered as those who completed the study, as inaction is a possible response to the intervention) | 3178 | 3198 | 3190
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline outcome measure was not applicable, since registration for vaccination was the outcome, and all participants were selected for not being registered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed Contact | Social Proof | Reframing Side Effects and Adverse Reactions | Total
Number analyzed (Participants) | 3178 | 3198 | 3190 | 9566
Age, Categorical [Count of Participants; unit: Participants] — Population: Data was not collected.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3178 | 3198 | 3190 | 9566

OUTCOME MEASURES:

1. Primary Outcome: Number of Employees Who Scheduled Vaccination Appointments After 3 Days
Description: Binary variable of a scheduled vaccination appointment 3 days after the emails were sent
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Contact | Social Proof | Reframing Side Effects and Adverse Reactions
Number analyzed (Participants) | 3178 | 3198 | 3190
Participants | 101 | 207 | 220
Statistical Analysis 1: Comparison: Delayed Contact vs Social Proof; We conducted a logistic regression with the two experimental conditions as dummy variables with delayed contact as the reference group; Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 2.11, 95% CI 2-sided [1.65 to 2.69]
Statistical Analysis 2: Comparison: Delayed Contact vs Reframing Side Effects and Adverse Reactions; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 2.26, 95% CI 2-sided [1.77 to 2.87]
Statistical Analysis 3: Comparison: Social Proof vs Reframing Side Effects and Adverse Reactions; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < .001, Regression, Logistic — We used an a priori threshold of p < .05; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.88 to 1.30]

2. Secondary Outcome: Number of Employees Who Opened Emails After 3 Days
Description: Binary variable indicating whether the employee opened the email 3 days after the emails were sent
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Social Proof | Reframing Side Effects and Adverse Reactions
Number analyzed (Participants) | 3198 | 3190
Participants | 1481 | 1398

3. Secondary Outcome: Number of Employees Who Clicked Scheduling Links After 3 Days
Description: Binary variable indicating whether the employee clicked the link to schedule a vaccination appointment 3 days after the emails were sent
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Social Proof | Reframing Side Effects and Adverse Reactions
Number analyzed (Participants) | 3198 | 3190
Participants | 562 | 382

4. Other Pre Specified Outcome: Number of Employees Who Scheduled Vaccination Appointments Until Policy Change (4 Days)
Description: Binary variable of a scheduled vaccination appointment up to the end of January 19, when new distribution policies were enacted.
Time Frame: 4 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Employees Who Opened Emails Until Policy Change (4 Days)
Description: Binary variable indicating whether the employee opened the email up to the end of January 19, when new distribution policies were enacted.
Time Frame: 4 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Employees Who Clicked the Scheduling Link Until Policy Change (4 Days)
Description: Binary variable indicating whether the employee clicked the link to schedule a vaccination appointment up to the end of January 19, when new distribution policies were enacted.
Time Frame: 4 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: No adverse events were evaluated.
Description: We only had access to email engagement data and registration data, which was kept separate from clinical data.
Arm/Group | Delayed Contact | Social Proof | Reframing Side Effects and Adverse Reactions
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
In the original ClinicalTrials record, the researchers preregistered that the study would examine primary and secondary outcomes after two days. This was extended to about three days, which was the time when the delayed control group was emailed. This altered timing was dictated by when the organization's marketing department was ready to send emails to the delayed control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT04728594/Prot_SAP_000.pdf